CLINICAL TRIAL: NCT06948669
Title: Predictors of Brain Death and Barriers to Organ Donation in a North African Intensive Care Units: A Multicenter Prospective Study on Severe Coma Patients
Brief Title: Brain Death and Organ Donation in Tunisian Intensive Care Units
Acronym: BDOD-TN
Status: Completed | Type: Observational
Sponsor: Faculty of Medicine, Sousse (Other)
Responsible Party: Principal Investigator, Imen Slama, Principal Investigator, Faculty of Medicine, Sousse
Other Study IDs: BDOD-Tunisia-2022-2023; HS13-2022 (Other: Sahloul University Hospital Research Ethics Committee)
Record Dates: First submitted 2025-04-11; First posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Brain Injury; Coma; Organ Transplants
Keywords: Organ donation refusal; ICU donor management; Cultural barriers; Hemorrhagic stroke outcome
MeSH Terms: conditions — Brain Injuries; Coma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study was to identify factors associated with the progression to brain death in critically ill patients with severe brain injuries in Tunisian intensive care units (ICUs). The main questions it aimed to answer were:

What medical factors (e.g., type of brain injury, ICU stay duration) increased the likelihood of progressing to brain death in these patients?

What patient characteristics (e.g., age, comorbidities) influenced the risk of brain death?

What were the reasons behind low organ donation rates in Tunisia, including family refusal and hospital-level barriers?

Participants were:

Adults with severe coma (Glasgow Coma Scale ≤ 8) requiring mechanical ventilation in Tunisian ICUs.

Data were collected as part of routine medical care, including information about medical factors, patient characteristics, and family attitudes towards organ donation, without any additional interventions beyond standard care.

The study was conducted from November 2022 to November 2023 across three ICUs: Sahloul, Farhat Hached, and Mohamed Taher Maamouri Hospitals.

DETAILED DESCRIPTION:
Background

Brain death (BD) is a legally and medically recognized condition under which organ donation may occur. However, organ donation rates in Tunisia remain low compared to international benchmarks. There is a need to better understand the factors influencing the progression to brain death in ICU patients, as well as the sociocultural and institutional barriers to organ donation in this setting.

Objectives

This study aimed to:

Identify clinical predictors of brain death among critically ill patients with severe brain injuries

Explore reasons for organ donation refusal by families

Identify hospital-level barriers in the organ donation process

Study Design and Setting

This was a prospective observational cohort study conducted between November 2022 and November 2023 in three Tunisian intensive care units:

Sahloul University Hospital (trauma center)

Farhat Hached University Hospital

Mohamed Taher Maamouri Hospital

Participants

Adult patients (≥18 years) admitted with severe coma (Glasgow Coma Scale ≤ 8) requiring mechanical ventilation were included. Patients with terminal illnesses unrelated to brain injury were excluded.

Procedures Data Collection

Data were prospectively collected using a standardized form developed and validated by experts in intensive care and the Tunisian National Centre for Organ Promotion and Transplantation (CNPTO).

The collected variables included:

Demographic information (e.g., age, sex)

Clinical characteristics (e.g., Glasgow Coma Scale on ICU admission, comorbidities, primary diagnosis)

Patient outcomes (e.g., progression to brain death, ICU discharge, or death from other causes)

Length of ICU stay

Organ donation process variables (e.g., whether families were approached, family consent or refusal, organ procurement, reasons for refusal)

Family approaches were conducted by the national transplant coordination team from the CNPTO.

No experimental interventions were applied. All procedures were part of standard ICU care.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years admitted to ICU with:

Severe coma (Glasgow Coma Scale ≤8)

Requiring mechanical ventilation

Primary diagnosis of:

Traumatic brain injury (TBI)

Hemorrhagic stroke

Other severe neurological conditions (anoxic brain injury, etc.)

Potential organ donor status (for brain death subgroup):

Meets clinical brain death criteria (absent brainstem reflexes, apnea)

Exclusion Criteria:

* Non-neurological terminal conditions: e.g., Advanced cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This prospective observational study enrolled 104 adult patients (≥18 years) with severe coma (Glasgow Coma Scale ≤8) requiring mechanical ventilation across three intensive care units in Tunisia.
  Key Features:
  Age/Sex: Mean age 47 years (range 18-80), 76% male
  Primary Conditions:
  Traumatic brain injury (61%)
  Hemorrhagic stroke (19%)
  Other neurological causes (20%)
  Study Groups:
  26 patients (25%) progressed to brain death
  78 patients (75%) did not
  Justification:
  The population represents typical severe coma cases in North African ICUs, with standardized brain death confirmation per national protocols (clinical exam + CT angiography).
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-25 (Actual)

PRIMARY OUTCOMES:
Brain death incidence | 0-12 months
  Proportion of patients progressing to brain death (clinical + CT angiography).
Family donation refusal rate | At time of brain death confirmation (through study completion, an average of 1 year)
  Percentage of families declining organ donation, with reasons

SECONDARY OUTCOMES:
Multivariate analysis of brain death predictors | From ICU admission to outcome determination (up to 1 year)
  Adjusted odds ratios (OR) for: 1) hemorrhagic stroke, 2) traumatic brain injury, and 3) ICU stay >14 days as independent predictors of brain death progression

CONTACTS AND LOCATIONS:
Overall Officials: Imed Chouchene, MD Professor, Study Director — Intensive Care Unit University Hospital of Farhat Hached Sousse Tunis Faculty of Medicine of Sousse
Locations (1):
- Faculty of Medicine of Sousse, University of Sousse, Sousse, Tunisia, Sousse, Tunisia

IPD SHARING:
Plan to Share IPD: No
No (but de-identified aggregate data will be published in the manuscript).

REFERENCES:
- [Derived] Slama I, Chouchene I, Ghammam R, Durin L, Naija W, Ziadi J, Ben Saad H. Predictors of brain death and barriers to organ donation in north African intensive care units: a multicenter prospective study on severe coma patients. Libyan J Med. 2025 Dec;20(1):2545049. doi: 10.1080/19932820.2025.2545049. Epub 2025 Aug 12. PMID 40794438